CLINICAL TRIAL: NCT05211479
Title: The Effect Of Tele-Nursing Application On Metabolic Control, Self-Efficacy, Quality Of Life And Anxiety Level Of Adolescents With Type 1 Diabetes
Brief Title: Tele Nursing Application For Type 1 Diabetes Mellitus Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Emel AVÇİN, Lecturer, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-14
Record Dates: First submitted 2021-11-25; First posted 2022-01-27 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Telenursing; Adolescent; Type 1 Diabetes Mellitus
Keywords: Telenursing; Type 1 Diabetes Mellitus; Metabolic Control; Self Efficacy; Quality of Life; Anxiety
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Anxiety Disorders | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Randomized controlled and quasi-experimental research
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Tele-nursing will be applied to adolescents in this group for 24 weeks. Weekly meeting and blood glucose monitoring will be done. The HbA1c value will be checked and the scales will be filled by meeting 3 times in total with 3 months intervals.
  Interventions: Behavioral: educational intervention
- Control Group (No Intervention): This group will be given face-to-face training only in the first encounter. During the research, no interviews will be provided through tele nursing. Only at the 3rd and 6th months will be interviewed to measure the HbA1c value and to fill the scales.

INTERVENTIONS:
Behavioral: educational intervention — In the light of up-to-date information, "Type I Diabetes Education Guide" was created. With this guide, both face-to-face and tele-nursing training will be provided. Both working groups will receive training before starting research. The intervention group will continue their weekly training throughout the study.
  Arms: intervention group

SUMMARY:
Studies have shown that tele-nursing practice is effective in children with Type 1 Diabetes Mellitus, but the number of studies conducted is very few. No study examining the concepts of metabolic control, self-efficacy, quality of life and anxiety together was found in the literature review. With this study, it is aimed that diabetes education given by tele-nursing has an effect on metabolic control, self-efficacy, quality of life and anxiety level of adolescents with type 1 diabetes, and that diabetic adolescents can easily obtain the information they need about nursing care when they cannot come to the clinic.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* The child is between the ages of 12-18,
* After the information, the adolescent agrees to participate in the study, and the parent gives written consent,
* The child can understand and speak Turkish,
* Parent's ability to understand and speak Turkish,
* Having a smart phone and having access to the internet,
* Having been diagnosed with T1DM at least 1 year ago,
* Being on insulin therapy by the subcutaneous route,
* Coming to the outpatient clinic at least once every 3 months.

Exclusion Criteria:

Exclusion Criteria:

* Age younger than 12 or older than 18,
* Having another chronic disease,
* Using an insulin pump
* Having vision and hearing problems,
* Using the Continuous Glucose Tracking System,
* Having a physical or mental disability.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of Metabolic control level of adolescents with type 1 diabetes | Baseline, 12 weeks and 24 weeks after randomization
  HbA1c values were recorded before starting the study to determine the level of metabolic control. The HbA1c values will be followed up in the 3rd and 6th months of the research. When the adolescents go to the hospital for a routine control every 3 months, the HbA1c value will be checked from the blood values and the researcher will obtain it from the records.
Evaluation of the level of self-efficacy of adolescents with type 1 diabetes | Baseline, 12 weeks and 24 weeks after randomization
  "Diabetes Self-Efficacy Scale in Adolescents with Type 1 Diabetes" was used to measure self-efficacy in diabetes management in adolescents aged 12-18 years with Type 1 Diabetes. Scale; medical treatment and nutrition, nutrition and insulin dose adjustment, being able to tell about diabetes, being honest with oneself and others (Ozturk, Ayar & Bektas, 2016). Participants will be asked to fill in the "Diabetes Self-Efficacy Scale in Adolescents with Type 1 Diabetes" scale to determine their self-efficacy levels in the 3rd and 6th months of the research.
Evaluation of the level of quality of life of adolescents with type 1 diabetes | Baseline, 12 weeks and 24 weeks after randomization
  "Quality of Life Scale for Children Adolescent Form (Kiddo-KINDL)" was used to determine the level of quality of life of adolescents. The scale form consists of 30 items and dimensions of physical well-being, mental well-being, self-esteem, family, friends, school, and illness (Eser et al., 2004). In the 3rd and 6th months of the study, participants will be asked to fill in the "Quality of Life Scale for Children Adolescent Form" scale to determine their quality of life.
Evaluation of the anxiety level of adolescents with type 1 diabetes | Baseline, 12 weeks and 24 weeks after randomization
  The scale is a self-report scale used in the evaluation of childhood anxiety disorders. The scale consists of 41 items and sub-dimensions of Panic Disorder/Somatic Disorder, Generalized Anxiety Disorder, Separation Anxiety, Social Anxiety, and School Fear. A cut-off value of 25 and above is accepted as a warning for anxiety disorder. An increase in the total score obtained from the scale means that the level of anxiety also increases (Cakmakcı, 2004). Participants will be asked to fill in the "Childhood Anxiety Screening Scale" scale to determine their anxiety levels in the 3rd and 6th months of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Emel AVÇİN, Doctorate, Principal Investigator — University of Yalova
Locations (1):
- Yalova University, Yalova, Turkey (Türkiye)

REFERENCES:
- [Derived] Avcin E, Acikgoz A. The effect of tele-nursing application on metabolic control, self-efficacy, quality of life and anxiety level in adolescents with Type 1 diabetes: A randomized controlled trial. J Pediatr Nurs. 2026 Feb 6;87:433-442. doi: 10.1016/j.pedn.2026.01.042. Online ahead of print. PMID 41653762